CLINICAL TRIAL: NCT05472870
Title: Efficacy and Mechanism of Repeated Transcranial Magnetic Stimulation in Children With Autism Spectrum Disorder: an Open-label Clinical Trial(Ⅱ)
Brief Title: Efficacy and Mechanism of rTMS in Children With ASD: an Open-label Clinical Trial(Ⅱ)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Fei Li, Chief Physician ,Doctoral Supervisor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2022-008-4
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Results first posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Repetitive Transcranial Magnetic Stimulation（rTMS）; Continuous theta Burst Stimulation （cTBS）
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- rTMS Group (Experimental): Participants will receive cTBS over the left primary motor cortext (M1) for 5 consecutive days. The detailed parameters as follows: 80% of RMT, 60 cycles of 10 bursts of three pulses at 50 Hz were delivered in 2-second trains (5 Hz) with no intertrain interval (i.e. triplet standard cTBS, 1800 pulses, 120s). Stimulation sessions were delivered hourly, 10 sessions were applied per day (18,000 pulses/day).
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — A technique that involves the use of electrical coils on the head to generate a brief magnetic field which reaches the cerebral cortex.

SUMMARY:
This study is a open-label clinical trial involving over 30 ASD children aged ≥4 years old. During the study, subjects received repeated transcranial magnetic stimulation (rTMS) intervention on the left primary motor cortex (M1) 10 times per day for 5 consecutive days and complete clinical assessments from pre-intervention to post-intervention. This study hopes to explore whether accelerated continuous theta-burst stimulation (a-cTBS) over left primary motor cortex (M1) can improve clinical symptoms of children with ASD in China.

DETAILED DESCRIPTION:
This study is a single-arm open-label clinical trial, designed to enroll at least 30 children with ASD aged over 4 years old.

During the trial, participants will receive accelerated continuous theta-burst stimulation (a-cTBS)on the left primary motor cortex (M1) for 5 consecutive days and complete clinical assessments within 2 weeks before the cTBS intervention (pre-cTBS), repeated within 3 days after the completion of the cTBS course (post-cTBS) and 1 month following the last cTBS session (one month follow-up), respectively. The purpose of this current study is to explore whether rTMS can improve the clinical symptoms of children with autism spectrum disorder in China, and to investigate the neurophysiological mechanism of rTMS for ASD children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged ≥4 years.
* Meeting the diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders, Edition 5 (DSM-5) .
* Confirmed by the ADOS and/or ADI-R diagnostic tool.
* Informed consent.

Exclusion Criteria:

* Patients with metal implants .
* Patients with neurological diseases such as epilepsy .
* Patients requiring surgical treatment due to structural abnormalities indicated by brain MRI .
* Genetic or chromosomal abnormalities .
* Suffering from mental disorders (such as mood disorders, etc.)
* Suffering from serious heart disease .
* Hearing-impaired .
* Intracranial hypertension .
* Participating in other clinical trials.
* Participants who received other interventions within 4 weeks prior to enrollment.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fei Li, Principal Investigator — Xinhua hospital Affilated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Fei Li, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- rTMS Group: Participants will receive accelerated continuous theta burst stimulation (a-cTBS, i.e. triplet standard cTBS, 1800 pulses/120s) for a 5 consecutive days, at an intensity that is 80% of the resting motor threshold (RMT) . a-cTBS repeats ten times a day with about 50 min interval . If feasible for the participant, all stimulation sessions will be held at the same time of the day. Treatment will be applied in left primary motor cortext (M1).
  repetitive Transcranial Magnetic Stimulation: A technique that involves the use of electrical coils on the head to generate a brief magnetic field which reaches the cerebral cortex.
Period: Overall Study
Arm/Group | rTMS Group
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- rTMS Group: Participants will receive accelerated continuous theta burst stimulation (a-cTBS, i.e. triplet standard cTBS, 1800 pulses/120s) for a 5 consecutive days, at an intensity that is 80% of the resting motor threshold (RMT) . a-cTBS repeats ten times a day with about 50 min interval . If feasible for the participant, all stimulation sessions will be held at the same time of the day. Treatment will be applied in left primary motor cortext (M1).
Arm/Group | rTMS Group
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.06 (1.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 30
Full Scale intelligence quotient (FSIQ) [Mean (Standard Deviation); unit: units on a scale] — We use the Wechsler Intelligence Scale to measure the intellectual ability of children. It can generate the full scale intelligence quotient (FSIQ) about children's the overall level of intelligence.
  The FSIQ ranges from 40-160, the higher values represent a better outcome.
  units on a scale | 74.97 (24.70)
Childhood Autism Rating Scale (CARS) [Mean (Standard Deviation); unit: units on a scale] — Childhood Autism Rating Scale (CARS) is one of the recommended diagnostic tools for ASD. It is comprised of 15 items (with a 4-point rating) covering a range of functions including social, emotional, adaptive, communicative, and cognitive.
  The CARS total score ranges from 15 to 60, a higher values represent a worse outcome.
  units on a scale | 33.48 (2.59)
Autism Diagnostic Observation Schedule (ADOS) [Mean (Standard Deviation); unit: units on a scale] — The Autism Diagnostic Observation Schedule (ADOS) is a standardized diagnostic test for assessing autism spectrum disorder. ADOS determined social, communication, and social-communication domains scores, here we use the social-communication domain score as the ADOS score(social score and communication score are summed to compute).
  ADOS score ranges from 0-20, a higher values represent a worse outcome.
  units on a scale | 13.73 (2.74)

OUTCOME MEASURES:

1. Primary Outcome: Social Response Scale (SRS) Scores
Description: Social Response Scale (SRS) is a parent questionnaire used to assess the presence and severity of social impairment. The SRS generates a total score and five subscale scores (social awareness, social cognition, social communication, social motivation, and autistic mannerisms), and 5 subscales scores are summed to compute the total score; higher scores indicate greater social impairment.
  The SRS total score range is "0-195", the social awareness subscale score range is "0-24", the social cognition subscale score range is "0-36", the social communication subscale score range is "0-66", the social motivation subscale score range is "0-33", and the autistic mannerisms subscale score range is "0-36".
  We collected the SRS from baseline to 1 month follow-up to evaluate the effect of rTMS treatment on ASD syptoms among these children.
Time Frame: Baseline, immediately after the completion of 5-days intervention, and 4 weeks after the completion of intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Group
Number analyzed (Participants) | 30
score on a scale
  Pre-intervention | 94.27 (20.26)
  Post-intervention | 81.50 (21.27)
  1month follow-up | 77.67 (20.13)
Statistical Analysis 1: Comparison: rTMS Group; All clinical behavioral data analysis was performed using Statistical Product and Service Solutions (SPSS) software (version 25.0). A P value <0.05 was considered statistically significant for all analyses. One-way ANOVA with repeated measures was used to examine differences in the effects of cTMS on the SRS; Test type: Superiority — One-way ANOVA with repeated measures was used to examine differences in the effects of cTMS on the SRS. A P value <0.05 was considered statistically significant for all analyses; p < 0.001, ANOVA — Bonferroni correction was used to adjust P values in post hoc analyses

2. Secondary Outcome: Childhood Autism Rating Scale (CARS)
Description: CARS is a behaviour-rating scale used to assess the presence and severity of the symptoms of autism spectrum disorder(ASD), with scores ranging from 15 to 60 and high scores indicating severe symptoms. Change of the CARS from baseline to 1 months after treatment to evaluate the effect of rTMS treatment on ASD.
  children.
Time Frame: Baseline, and 4 weeks after the completion of intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Group
Number analyzed (Participants) | 30
score on a scale
  pre-intervention | 33.48 (2.59)
  1month follow-up | 32.83 (2.66)

3. Secondary Outcome: Behavior Rating Inventory of Executive Function (BRIEF)
Description: BRIEF is a quick and efficient measure of executive function(have school-age version (BRIEF-S) and preschool version (BRIEF-P)), we asked parents to complete the 86-item (BRIEF-S) or 63-item (BRIEF-P) form to rate a child's executive functions (1-3 score) within the context of his everyday environments (home or school).
  Here we report the BRIEF composite score, BRIEF-S score range is 86 -258 and BRIEF-P score range is 63-189. The higer scores indicate more impairment in executive function.
  We evaluate the changes in executive function (EF) scores before and after cTBS treatment.
Time Frame: Baseline, immediately after the completion of 5-days intervention, and 4 weeks after the completion of intervention.
Population: Three parents of participants did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- rTMS Group (School Age): Participants will receive accelerated continuous theta burst stimulation (a-cTBS, i.e. triplet standard cTBS, 1800 pulses/120s) for a 5 consecutive days, at an intensity that is 80% of the resting motor threshold (RMT) . a-cTBS repeats ten times a day with about 50 min interval . If feasible for the participant, all stimulation sessions will be held at the same time of the day. Treatment will be applied in left primary motor cortext (M1).
  Children who are already in school need to complete the school-age version
- rTMS Group (Preschool Age): Participants will receive accelerated continuous theta burst stimulation (a-cTBS, i.e. triplet standard cTBS, 1800 pulses/120s) for a 5 consecutive days, at an intensity that is 80% of the resting motor threshold (RMT) . a-cTBS repeats ten times a day with about 50 min interval . If feasible for the participant, all stimulation sessions will be held at the same time of the day. Treatment will be applied in left primary motor cortext (M1).
  Children who are not yet in school need to complete the preschool-age version
Arm/Group | rTMS Group (School Age) | rTMS Group (Preschool Age)
Number analyzed (Participants) | 17 | 10
score on a scale
  Pre-intervention | 153.76 (20.55) | 115.30 (10.09)
  Post-intervention | 152.76 (20.28) | 117.60 (14.24)
  1month follow-up | 149.12 (18.35) | 112.00 (10.59)

4. Secondary Outcome: Conners Parent Symptom Questionnaire (PSQ)
Description: Conners Parent Symptom Questionnaire (PSQ) is a questionnaire screening for children's behavioral problems (especially with ADHD), it has 48 items（4-stage: 0-3) that can be divided into 6 factors (conduct problems, learning problems, psychosomatic problems, impulsive-hyperactivity, anxiety, and hyperactivity index). Add the scores and divide by the item numbers of each factor to get Z score.
  Here we mainly observe the changes in Hyperactivity Index (HI) Z scores, it ranges from 0-3, a higher score mean a worse outcome.
Time Frame: Baseline, immediately after the completion of 5-days intervention, and 4 weeks after the completion of intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Group
Number analyzed (Participants) | 30
score on a scale
  Pre-intervention | 1.20 (0.49)
  Post-intervention | 1.18 (0.48)
  1month follow-up | 1.10 (0.34)

5. Secondary Outcome: Peabody Picture Vocabulary Test（PPVT）
Description: The Peabody Picture Vocabulary Test is one of the most commonly used assessment tests for measuring single-word comprehension. The raw score ranges from 0-110, the higher scores mean a better outcome. we collected the PPVT raw score from baseline to 1 months after treatment to evaluate the effect of rTMS treatment on ASD children's words comprehension.
Time Frame: Baseline, and 4 weeks after the completion of intervention.
Population: Three subjects did not cooperate with the test, so their data were excluded from the analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Group
Number analyzed (Participants) | 27
score on a scale
  Pre-intervention | 67.78 (27.23)
  1month follow-up | 76.11 (26.89)

6. Secondary Outcome: Chinese Communicative Development Inventory (CCDI)
Description: CCDI provides a powerful tool to assess early vocabulary development and the language skills of older children with developmental disorders and the effectiveness of their intervention. Here we collected the CCDI words produced score, it ranges from 0-798. The higher scores mean a better outcome.
Time Frame: Baseline and 4 weeks after the completion of intervention.
Population: 8 subjects whose parents did not complete the follow-up scale or who had reached the highest measurable score on the scale in terms of ability (ceiling effect) were not included in the analysis
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | rTMS Group
Number analyzed (Participants) | 22
score on a scale
  Pre-intervention | 733.00 [615.25 to 789.50]
  1month follow-up | 771.50 [657.00 to 793.25]

7. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I)
Description: CGI is a scale used to assess the severity of the illness and the global improvement of the patient under intervention. Here we used Clinical Global Impression of Improvement (CGI-I) to rate how much the patient's illness has improved or worsened relative to baseline (a seven-point scale: 1 = "very much improved" to 7 = "very much worse"). The CGI was carried out by trained clinical assessors according to children's CARS、ADOS assessment results and parent interviews before and after intervention. We calculated the number of subjects with improvement (CGI-I≤3).
Time Frame: After the completion of 5-days intervention and 4 weeks after the completion of intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | rTMS Group
Number analyzed (Participants) | 30
Participants
  Post-intervention | 20
  1month follow-up | 27

8. Secondary Outcome: Repetitive Behaviors Scale - Revised (RBS-R)
Description: The Repetitive Behaviors Scale - Revised (RBS-R) is a 44-item (rated 0-3) questionnaire that is used to measure the breadth of repetitive behavior in children, adolescents, and adults with Autism Spectrum disorders. The RBS-R provides a quantitative, continuous measure of the full spectrum of repetitive behaviors. The RBS-R consists of six subscales including: Stereotyped Behavior, Self-injurious Behavior, Compulsive Behavior, Routine Behavior, Sameness Behavior, and Restricted Behavior, that have no overlap of item content.
  Here we use the RBS-R total score, it ranges from 0-132, the higher score means worse repetitive behavior.
Time Frame: baseline, immediately after the completion of 5-days intervention, and 4 weeks after the completion of intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | rTMS Group
Number analyzed (Participants) | 30
score on a scale
  Pre-intervention | 7.00 [4.75 to 9.00]
  immediately after the completion of Post-intervention | 7.00 [4.75 to 9.00]
  4 weeks after the completion of 1month follow-up | 5.5 [3.75 to 8.00]

9. Other Pre Specified Outcome: Power Spectral Density (PSD) Within the Alpha Frequency Band
Description: For EEG data, we caculated the power spectral density (PSD) within the alpha frequency band (8-13 Hz) for all channels.
Time Frame: Baseline, immediately after the completion of 5-days intervention.
Population: We successfully collected EEG data from 26 children before and after the intervention, and one patient was excluded after a quality control procedure. Due to limited implementation conditions (e.g., epidemics, installations) , we did not collect EEG data at 1-month follow-up. The phase locking value(PLV) and coherence (Coh) were not analyzed due to data and analyst issues.
Measure: Mean (Standard Deviation); unit: W/Hz
Arm/Group | rTMS Group
Number analyzed (Participants) | 25
W/Hz
  Pre-intervention | 2.05 (0.96)
  Post-intervention | 1.66 (0.67)

10. Other Pre Specified Outcome: Multilingual Assessment Instrument for Narratives (MAIN)
Description: For a subset of ASD children with adequate expressive ability (those able to at least use phrases), we use Multilingual Assessment Instrument for Narratives (MAIN) tool to assess their narrative comprehension and production skills. In this test, children were asked to tell and retell the story and answer comprehension questions, and then assessors scored children's performance from four dimensions (i.e., story structure, structural complexity, and internal state terms and comprehension questions). The story structure score range is 0-18, structural complexity score range is 0-4, internal state terms score range is 0-no limit, and comprehension questions score range is 0-10. The higher score means better performance.
Time Frame: Baseline, and 4 weeks after the completion of intervention.
Population: 14 children having certain expression ability to complete MAIN test.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | rTMS Group
Number analyzed (Participants) | 14
score on a scale
  Telling_Story Structure_Pre-intervention | 7.57 (2.34)
  Telling_Story Structure_1month follow-up | 8.96 (2.43)
  Telling_Structural Complexity_Pre-intervention | 2.11 (0.59)
  Telling_Structural Complexity_1month follow-up | 2.50 (0.55)
  Telling_Internal States Terms_Pre-intervention | 3.68 (2.00)
  Telling_Internal States Terms_1month follow-up | 5.21 (3.20)
  Telling_Comprehension Questions_Pre-intervention | 6.50 (1.79)
  Telling_Comprehension Questions_1month follow-up | 8.32 (1.56)
  Retelling_Story Structure_Pre-intervention | 9.07 (2.18)
  Retelling_Story Structure_1month follow-up | 12.21 (2.28)
  Retelling_Structural Complexity_Pre-intervention | 2.32 (0.58)
  Retelling_Structural Complexity_1month follow-up | 2.75 (0.38)
  Retelling_Internal States Terms_Pre-intervention | 5.07 (2.13)
  Retelling_Internal States Terms_1month follow-up | 6.14 (1.56)
  Retelling_Comprehension Questions_Pre-intervention | 6.46 (1.96)
  Retelling_Comprehension Questions_1month follow-up | 8.21 (1.66)

ADVERSE EVENTS:
Time Frame: A semi-structured interview was administered following each treatment session and 1 month follow-up.
Description: rating the event as mild (no impairment, no need stopping trial), moderate (some impairment, need stopping trial, no need for intervention), severe (evidence of impairment, need stopping trial and need for intervention).
Arm/Group | rTMS Group
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 8/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rTMS Group (N=30)
agitation (Nervous system disorders) | 6 — during intervention period, mild and disappeared without any specific therapy.
scalp pain (Skin and subcutaneous tissue disorders) | 3 — during the first few stimulation treatments, mild and disappeared without any specific therapy.
nausea (Nervous system disorders) | 1 — Occurred once during the follow-up period after full-doses treatment, disappeared without any specific therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT05472870/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05472870/ICF_001.pdf